CLINICAL TRIAL: NCT04669392
Title: Clinical and Radiographic Evaluation of 70% Ethanol Alcohol Versus Normal Saline as Root Canal Irrigating Solutions in Partial Pulpectomy of Primary Molars With Metapex A Randomized Controlled (Pilot Trial)
Brief Title: The Effect of Using 70% Ethanol Alcohol as a Root Canal Irrigant on Increasing the Success Rate of Metapex in Pulpectomy Compared to Normal Saline in Primary Molars
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Thamar Al-Gannah Samy Rashed, Thamar Al-Gannah Samy Mohamed Rashed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12021
Record Dates: First submitted 2020-12-12; First posted 2020-12-16 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Pulpitis - Irreversible; Resorption, Root; Abscess Bone; Mobility, Tooth; Pain
Keywords: Metapex; Primary dentition
MeSH Terms: conditions — Root Resorption; Tooth Mobility; Pain | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 70% Ethanol (Experimental): Using 70% Ethanol Alcohol as a root canal irrigating solution before obturating the lower primary second molar with Metapex
  Interventions: Drug: 70% Ethanol Alcohol
- Normal Saline (No Intervention): Irrigating the canals with Normal Saline before obturating the lower primary second molar with Metapex

INTERVENTIONS:
Drug: 70% Ethanol Alcohol — Ethanol, also called ethyl alcohol, grain alcohol, or alcohol, a member of a class of organic compounds that are given the general name alcohols.
  Ethanol is a commonly used fixative. Fixation of the inner layers of the tissue depends on the ability of the fixative to diffuse into the tissue. Moreover, Ethanol has antibacterial antifungal, and antiviral properties.
  70% Ethanol is the safest concentration because the water that has been mixed into the ethanol slows the drying time, creating a longer contact time. Ethanol needs to have a contact time of at least 10 seconds to kill Staphylococcus aureus and Streptococcus pyogenes. At a 10 second drying time.
  Arms: 70% Ethanol

SUMMARY:
The aim of the study is to perform a clinical and radiographic evaluation of 70% Ethanol Alcohol versus Normal Saline as root canal irrigating solutions in partial pulpectomy of primary molars with Metapex.

DETAILED DESCRIPTION:
In permanent dentition, Calcium Hydroxide-Iodoform paste (Metapex) has a high potential in forming a calcific barrier in the pulpal tissue. Yet, in primary dentition Metapex forms a chronic inflammatory reaction to the pulpal tissue leading to its internal and root resorption. Although the high success rate of Metapex in partial pulpectomy, the rapid resorption of Metapex has led to the presence of the hollow tube effect due to voids formation in the canals. However, this will cause early root resorption before the time of exfoliation. Due to its rapid resorption, Metapex is usually recommended to be used in the pulpectomy of teeth near exfoliation in order to avoid the early root resorption of primary dentition in order to avoid the premature loss of the endodontically treated vital primary teeth with Metapex.

Saline solution is the basic irrigating solution in root canal treatments, yet it has no antimicrobial activities and only results in cleaning the root canals. Ethanol irrigation is believed to be an alternative promising replacement in tissue fixation from Formocresol due to the concerns from its carcinogenicity and toxicity. Also, Ethanol has an excellent bactericidal, virucidal, and fungicidal, and most importantly it is one of the volatile liquids.

In this study, the effect of Ethanol Alcohol on increasing the success rate of Metapex in vital pulp therapy will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients medically within normal.
2. Cooperative patients and cooperative parents.
3. Children aged 4-7 years old.
4. Primary mandibular second molar.
5. Deep carious molars.
6. A history of spontaneous pain.
7. Molars with pulp exposure due to caries.
8. Absences of Internal resorption.
9. Absences of external pathological resorption.
10. where the bleeding could not be stopped following removal of the coronal pulp tissue

Exclusion Criteria:

1. Parents unable to give informed consent.
2. Necrotic pulp.
3. Unrestorable Teeth.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain of partial pulpectomy of Metapex using both 70% Ethanol Alcohol and Normal Saline as root canal irrigating solutions. | Patients will be assessed at 12 months follow ups
  Assessment through Visual Analog Scale , A score from (0-10) 0 is means no pain and 10 is the maximum level of pain.

SECONDARY OUTCOMES:
Radiographic evaluation of partial pulpectomy of Metapex using both 70% Ethanol Alcohol and Normal Saline as root canal irrigating solutions. | Patients will be assessed at 12 months follow ups
  Assessment through Visual interpretation of digital radiograph

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brand, C. & At, D. M. E. Guidelines for Disinfection and Sterilization in Healthcare Facilities , 2008 ( Centers for Disease Control ). 2008, (2008).
- [Result] Nurko C, Ranly DM, Garcia-Godoy F, Lakshmyya KN. Resorption of a calcium hydroxide/iodoform paste (Vitapex) in root canal therapy for primary teeth: a case report. Pediatr Dent. 2000 Nov-Dec;22(6):517-20. PMID 11132515
- [Result] Al-Ostwani AO, Al-Monaqel BM, Al-Tinawi MK. A clinical and radiographic study of four different root canal fillings in primary molars. J Indian Soc Pedod Prev Dent. 2016 Jan-Mar;34(1):55-9. doi: 10.4103/0970-4388.175515. PMID 26838149
- [Result] Thiruvenkadam G, Asokan S, John B, Priya PG. Effect of 95% Ethanol as a Final Irrigant before Root Canal Obturation in Primary Teeth: An in vitro Study. Int J Clin Pediatr Dent. 2016 Jan-Mar;9(1):21-4. doi: 10.5005/jp-journals-10005-1327. Epub 2016 Apr 22. PMID 27274150
- [Result] Panzacchi S, Gnudi F, Mandrioli D, Montella R, Strollo V, Merrick BA, Belpoggi F, Tibaldi E. Effects of short and long-term alcohol-based fixation on Sprague-Dawley rat tissue morphology, protein and nucleic acid preservation. Acta Histochem. 2019 Aug;121(6):750-760. doi: 10.1016/j.acthis.2019.05.011. Epub 2019 Jul 3. PMID 31277893